CLINICAL TRIAL: NCT04411953
Title: A Single Center, Single Dose, Open-label, Randomized, Two Period Crossover Pivotal Study to Determine the Bioequivalence of Two Formulations Containing Haloperidol 2 mg in Healthy Males and Females Under Fed Conditions
Brief Title: Bioequivalence Study of Two Oral Haloperidol Tablets Formulations in Healthy Subjects Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cycle Pharmaceuticals Ltd. (Industry)
Collaborators: Farmovs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CT-006; 0145FRM18 (Other: FARMOVS Clinical Research Organisation)
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-03

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Benztropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference Product (Treatment A) (Active Comparator): Subjects received Haloperidol Tablets 2 mg Reference Product (Mylan Pharmaceuticals Inc.). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Interventions: Drug: Haloperidol Tablets, Mylan Pharmaceuticals Inc.
- Test Product (Treatment B) (Experimental): Subjects received Haloperidol Tablets 2 mg Test Product (Cycle Pharmaceuticals Ltd). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Interventions: Drug: Haloperidol Tablets, Cycle Pharmaceuticals Ltd

INTERVENTIONS:
Drug: Haloperidol Tablets, Mylan Pharmaceuticals Inc. — single dose, 2 mg Haloperidol tablet
  Other Names: Benztropine Mesylate Tablets
  Arms: Reference Product (Treatment A)
Drug: Haloperidol Tablets, Cycle Pharmaceuticals Ltd — single dose, 2 mg Haloperidol tablet
  Other Names: Benztropine Mesylate Tablets
  Arms: Test Product (Treatment B)

SUMMARY:
The purpose on this study was to determine whether the test product, Haloperidol Tablets, 2 mg (Cycle Pharmaceuticals Ltd), and the reference product, Haloperidol Tablets, United States Pharmacopeia (USP), 2 mg (Mylan Pharmaceuticals Inc.) are bioequivalent under fed conditions.

DETAILED DESCRIPTION:
The specific aim was to conduct a single dose, open-label, randomized, two period crossover pivotal study to determine the bioequivalence of two formulations containing haloperidol 2 mg in healthy males and females under fed conditions.

A total of 32 healthy female and male volunteers (age 18 to 55 years old) were entered into the study. Volunteers were determined to be free of significant medical conditions as assessed by medical history, physical examination, and blood and urine tests. Volunteers were randomly allocated to a treatment sequence, before administration of investigational medicinal product (IMP) under fed conditions.

A wash-out period of at least 14 calendar days (minimum number of days based on half-life of the analyte) between consecutive administrations of the IMP was maintained.

Blood samples were collected at at pre-dose (0 hours), at 30 minutes, at 1 hour,

1 hour 30 minutes, 2 hours, 2 hours 30 minutes, 3 hours, 3 hours 30 minutes, 4 hours, 4 hours 30 minutes, 5 hours, 5 hours 30 minutes, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours, 168 hours and 192 hours post-dose (total: 26 samples per treatment period).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 30 kg/m^2 (both inclusive).
* Body mass not less than 50 kg.
* Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the investigator considers the deviation to be irrelevant for the purpose of the study.
* Non-smokers.
* Females, if:
* Not of childbearing potential, e.g., has been surgically sterilized, undergone a hysterectomy, amenorrhea for ≥ 12 months and considered post-menopausal, Note: In post-menopausal women, the value of the serum pregnancy test may be slightly increased. This test will be repeated to confirm the results. If there is no increase indicative of pregnancy, the female will be included in the study.
* Of childbearing potential, the following conditions are to be met:
* Negative pregnancy test If this test is positive, the subject will be excluded from the study. In the rare circumstance that a pregnancy is discovered after the subject received IMP, every attempt must be made to follow her to term.
* Not lactating
* Abstaining from sexual activity (if this is the usual lifestyle of the subject) or must agree to use an accepted method of contraception, and agree to continue with the same method throughout the study An example of a reliable method of contraception is a non-hormonal intrauterine device. In this study the concomitant use of hormonal contraceptives is NOT allowed. Other methods, if considered by the investigator as reliable, will be accepted.
* Written consent given for participation in the study.
* Written consent given for participation in the genetic component of the study (if performed based on Food and Drug Administration (FDA) feedback). If the subject declines participation in the genetic component, the subject will not be allowed to participate in the study.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females (1 unit is equal to approximately 330 mL of beer, one small glass [200 mL] of wine, or one measure [25 mL] of spirits).
* Regular exposure to substances of abuse (other than alcohol) within the past year.
* Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks before the first administration of IMP except if this will not affect the outcome of the study in the opinion of the investigator. In this study the concomitant use of hormonal contraceptives is NOT allowed.
* Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks (or within 5 elimination half-lives for chemical entities or 2 elimination half-lives for antibodies or insulin, whichever is the longer) before administration of IMP in this study, at the discretion of the investigator.
* Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
* A major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity or allergy to the IMP or its excipients or any related medication.
* History of hypersensitivity or allergy to the pre-medication or its excipients or any related medication.
* History of hypersensitivity or allergy to the rescue medication or its excipients or any related medication.
* History of bronchial asthma or any other bronchospastic disease.
* History of convulsions.
* History of porphyria.
* History of cardiac arrhythmias.
* History of sudden cardiac death in the family or history of familial long QT syndrome.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Cytochrome P450 (CYP) 2D6 poor metabolizers (if warranted by the FDA).
* Hypomagnesemia.
* Hypothyroidism or hyperthyroidism.
* Hypokalemia.
* Subjects with narrow-angle glaucoma.
* Subjects with stenosing peptic ulcers.
* Subjects who have pyloroduodenal obstruction.
* Subjects who have symptomatic prostatic hypertrophy or bladder-neck obstruction.
* Known or previous dystonia or dyskinesia.
* Subjects with severe toxic central nervous system depression or who have experienced comatose states from any cause.
* Subjects who have Parkinson's disease.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP.
* Diagnosis of hypotension made during the screening period.
* Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
* Positive testing for human immunodeficiency virus (HIV), hepatitis B and hepatitis C.
* Positive urine screen for drugs of abuse. In case of a positive result the urine screen for drugs of abuse may be repeated once at the discretion of the investigator.
* Positive pregnancy test (female subjects).
* Hemoglobin count deviating more than 10% of the lower limit of normal.
* Veins unsuitable for venous blood collection.
* Difficulty in swallowing.
* Any specific IMP safety concern.
* Vulnerable subjects, e.g., persons in detention.
* Employees or close relatives of the contract research organization, the sponsor, 3rd party vendors or affiliates of the above mentioned parties.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- FARMOVS Clinical Research Organisation, Bloemfontein, Free State, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 subjects participated in the screening phase of this study.
Pre-assignment Details: 32 subjects were enrolled in the study. 24 subjects were excluded from the study. 3 subjects were placed on standby.
Groups:
- Reference Product (Treatment A), Then Test Product (Treatment B): Treatment A: Subjects received Haloperidol Tablets 2 mg Reference Product (Mylan Pharmaceuticals Inc.). Subjects also received as pre-medication Benztropine Mesylate Tablets, United States Pharmacopeia (USP) (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with Investigational Medicinal Product (IMP) and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Haloperidol Tablets, Mylan Pharmaceuticals Inc.: single dose, 2 mg Haloperidol tablet
  Then
  Treatment B:
- Test Product (Treatment B), Then Reference Product (Treatment A): Treatment B: Subjects received Haloperidol Tablets 2 mg Test Product (Cycle Pharmaceuticals Ltd). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Haloperidol Tablets, Cycle Pharmaceuticals Ltd: single dose, 2 mg Haloperidol tablet
  Then
  Treatment A: Subjects received Haloperidol Tablets 2 mg Reference Product (Mylan Pharmaceuticals Inc.). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
Period: Treatment Period 1 (8 Days)
Arm/Group | Reference Product (Treatment A), Then Test Product (Treatment B) | Test Product (Treatment B), Then Reference Product (Treatment A)
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout Period (14 Days)
Arm/Group | Reference Product (Treatment A), Then Test Product (Treatment B) | Test Product (Treatment B), Then Reference Product (Treatment A)
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1
Period: Treatment Period 2 (8 Days)
Arm/Group | Reference Product (Treatment A), Then Test Product (Treatment B) | Test Product (Treatment B), Then Reference Product (Treatment A)
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence AB: Treatment A: Subjects received Haloperidol Tablets 2 mg Reference Product (Mylan Pharmaceuticals Inc.). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Haloperidol Tablets, Mylan Pharmaceuticals Inc.: single dose, 2 mg Haloperidol tablet
  Treatment B: Subjects received Haloperidol Tablets 2 mg Test Product (Cycle Pharmaceuticals Ltd). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Haloperidol Tablets, Cycle Pharmaceuticals Ltd: single dose, 2 mg Haloperidol tablet
- Sequence BA: Treatment B: Subjects received Haloperidol Tablets 2 mg Test Product (Cycle Pharmaceuticals Ltd). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Haloperidol Tablets, Cycle Pharmaceuticals Ltd: single dose, 2 mg Haloperidol tablet
  Treatment A: Subjects received Haloperidol Tablets 2 mg Reference Product (Mylan Pharmaceuticals Inc.). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Haloperidol Tablets, Mylan Pharmaceuticals Inc.: single dose, 2 mg Haloperidol tablet
- Total: Total of all reporting groups
Arm/Group | Sequence AB | Sequence BA | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.3 (9.64) | 26.2 (6.30) | 27.3 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 12 | 15 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 1 | 2 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 16 | 16 | 32
Height [Mean (Standard Deviation); unit: cm] | 170.53 (8.586) | 168.64 (8.380) | 169.59 (8.401)
Weight [Mean (Standard Deviation); unit: kg] | 69.69 (12.121) | 65.63 (10.036) | 67.66 (11.139)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.90 (3.300) | 23.03 (2.763) | 23.47 (3.026)

OUTCOME MEASURES:

1. Primary Outcome: Concentration Maximum (Cmax)
Description: The maximum observed concentration of haloperidol as measured by bioanalysis of the blood plasma is referred to as the Cmax.
Time Frame: pre-dose (0 hours), and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144, 168, 192 hours post dose
Population: One subject was withdrawn after the interim safety analysis during the washout period and so did not complete Treatment Period 2 (the subject was scheduled to receive Test Product (Treatment B)). Since only 31 subjects completed the study, only 31 subjects were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Reference Product (Treatment A): Subjects received Haloperidol Tablets 2 mg Reference Product (Mylan Pharmaceuticals Inc.). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Haloperidol Tablets, Mylan Pharmaceuticals Inc.: single dose, 2 mg Haloperidol tablet
- Test Product (Treatment B): Subjects received Haloperidol Tablets 2 mg Test Product (Cycle Pharmaceuticals Ltd). Subjects also received as pre-medication Benztropine Mesylate Tablets, USP (1 mg every 10 to 12 hours), beginning 4 to 6 hours before dosing with IMP and continued for a total of 4 doses.
  A high-fat, high-calorie breakfast was served 30 minute before administration of the IMP.
  Haloperidol Tablets, Cycle Pharmaceuticals Ltd: single dose, 2 mg Haloperidol tablet
Arm/Group | Reference Product (Treatment A) | Test Product (Treatment B)
Number analyzed (Participants) | 31 | 31
ng/ml | 1.326 (0.4338) | 1.293 (0.3919)

2. Primary Outcome: Area Under the Curve (0-t) (AUC(0-t))
Description: Area under the plasma concentration versus time curve from time zero to t, where t is the time of the timepoint of the last quantifiable concentration of haloperidol in the blood plasma. The curve is constructed by plotting the concentration of haloperidol in the blood plasma against the time for each blood sample.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Reference Product (Treatment A) | Test Product (Treatment B)
Number analyzed (Participants) | 31 | 31
h*ng/ml | 27.75 (10.19) | 28.46 (11.78)

3. Primary Outcome: Area Under the Curve(0-∞) (AUC(0-∞))
Description: Area under the plasma concentration versus time curve from time zero to ∞, where ∞ is the timepoint of the last quantifiable concentration of haloperidol in the blood plasma, plus it's elimination rate constant. AUC(0-∞) = AUC(0-t) + AUC(t-∞).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Reference Product (Treatment A) | Test Product (Treatment B)
Number analyzed (Participants) | 31 | 31
h*ng/ml | 30.61 (11.29) | 31.34 (12.06)

4. Secondary Outcome: Time to Maximum Concentration (Tmax)
Description: The timepoint at which the maximum concentration of haloperidol as measured by bioanalysis of the blood plasma is observed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Reference Product (Treatment A) | Test Product (Treatment B)
Number analyzed (Participants) | 31 | 31
Hours | 4.871 (3.750) | 3.839 (1.274)

5. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Description: Terminal elimination rate constant (λz) is a mathematical estimate calculated using log-linear regression of the terminal portions of a blood plasma concentration against time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Reference Product (Treatment A) | Test Product (Treatment B)
Number analyzed (Participants) | 31 | 31
1/h | 0.01114 (0.003451) | 0.01152 (0.004028)

6. Secondary Outcome: Terminal Elimination Half-life (t½)
Description: The apparent terminal elimination half-life (t½) is defined as the time necessary for the concentration of a drug to decrease by one-half in the terminal phase.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Reference Product (Treatment A) | Test Product (Treatment B)
Number analyzed (Participants) | 31 | 31
Hours | 69.12 (26.40) | 70.19 (35.25)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected for the duration of the study (24 days).
Arm/Group | Reference Product (Treatment A) | Test Product (Treatment B)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 21/31 | 21/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference Product (Treatment A) (N=31) | Test Product (Treatment B) (N=32)
Dry Mouth (Gastrointestinal disorders) | 6 (7) | 7 (8)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 5 (5)
Headache (Nervous system disorders) | 4 (6) | 2 (2)
Vision Blurred (Eye disorders) | 4 (4) | 5 (5)
Eye Pruritus (Eye disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Non-cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Hypervigilance (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT04411953/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT04411953/SAP_001.pdf